CLINICAL TRIAL: NCT06376032
Title: EndeavorOTC® Research Study in College Students
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akili Interactive Labs, Inc. (Industry)
Collaborators: Landmark College (Unknown); Villa Maria College (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Akili-068
Record Dates: First submitted 2024-04-17; First posted 2024-04-19 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Attention; Cognition; University Students

STUDY DESIGN:
Intervention Model Description: Eligible students will be randomized* to two cohorts: the first will receive immediate access to AKL-T01, and the second will complete weekly online surveys and receive access to AKL-T01 after the first group has completed the recommended 6 weeks of use. Regardless of group assignment, all participants will receive full 12-weeks of access to AKL-T01 during the course of the study.
  *Depending on enrollment numbers for a given semester (e.g., if <100 students are enrolled and the study is underpowered to conduct between-group comparisons), all participants may be assigned to receive treatment immediately (i.e., single-arm design) and primary study hypotheses may be evaluated according to within-person changes in outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Group 1 (Experimental): Participants receive immediate 12-week access to EndeavorOTC.
  Interventions: Device: EndeavorOTC®
- Group 2 (Experimental): Participants receive 12-week access to EndeavorOTC 6-weeks after Group 1.
  Interventions: Device: EndeavorOTC®

INTERVENTIONS:
Device: EndeavorOTC® — EndeavorOTC is an over the counter digital therapeutic designed to improve attention function as measured by computer-based testing in patients 18 and older with primarily inattentive or combined type ADHD, who have a demonstrated attention issue. EndeavorOTC utilizes the same proprietary technology underlying EndeavorRx®, an FDA-authorized prescription digital therapeutic indicated to improve attention function in children ages 8-17. EndeavorOTC is deployed on mobile devices and incorporates adaptive, simultaneous cognitive tasks in a consumer-grade action videogame-based platform with high-quality graphics and reward mechanisms.
  Other Names: AKL-T01A

SUMMARY:
The objective of this study is to evaluate the impact of a digital therapeutic (EndeavorOTC®, also known as AKL-T01A) on clinical symptoms of executive and cognitive functioning in a real-world sample of university students. This study aims to answer whether EndeavorOTC represents a useful intervention for targeting broad cognitive and emotional health among university students.

DETAILED DESCRIPTION:
University students face an increased risk of mental health challenges, as well as elevated stress due to the demands of managing coursework and social stress during a formative developmental period with increased independence. Consequently, there is a need for scalable, evidence-based interventions that can help university students manage their cognitive and emotional health. Through a partnership between Akili Interactive Labs and participating colleges, free 12-week access to AKL-T01 will be provided to any student interested in treatment for the duration of an academic semester, up to an N of 500 per site. This study will evaluate changes in participants across a range of clinical and functional outcomes, including cognitive functioning, academic outcomes, social functioning, attention and associated symptoms, and quality of life. The study will also evaluate user feedback and information on the usability of AKL-T01 through both quantitative and qualitative methods.

ELIGIBILITY:
Inclusion Criteria:

* Owns a personal Android or iOS device to access AKL-T01 treatment
* Provides informed consent to participate in this study
* Is 18 years of age or older

Exclusion Criteria:

* Known photosensitive epilepsy, color blindness, and any physical limitation that would make engagement with an app-based digital intervention difficult
* Has participated in the same study in previous semesters

Pregnant and nursing people are eligible to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Computerized Adaptive Test, Mental Health (CAT-MH®) | Baseline, Exit (Day 84)
  Computerized Adaptive Test, Mental Health (CAT-MH®) is a distinct suite of computer adaptive tests that is based on multidimensional item response theory. The adult ADHD module is a dimensional severity measure of attention-deficit/hyperactivity disorder symptomatology for adults 18 and over. The number and selection of questions within the assessment varies as individuals' initial item responses are used to determine a provisional estimate of their standing on the measured trait to be used for subsequent item selection. Items are scored on a Likert scale of 1 (Not at all), 2 (Just a little), 3 (Somewhat), 4 (Quite a bit), and 5 (Very much).
  Negative change in score indicates improvement in ADHD severity.
PROMIS Cognitive Function v2.0 - Short Form | Baseline, Day 42, Day 84
  The PROMIS Cognitive Function v2.0 short form consists of six questions about the respondent's cognitive function in the past 7 days rated on a Likert scale of 1-5, where 1=Very often (Several times a day) and 5=Never.
  Higher score indicates higher levels of cognition. Positive change in score indicates improvement.
PROMIS Satisfaction with Participation in Discretionary Social Activities (v1.0) | Baseline, Day 42, Day 84
  The PROMIS Satisfaction with Participation in Discretionary Social Activities scale consists of 7 questions about the respondent's satisfaction in the past 7 days rated on a Likert scale of 1-5 where 1=Not at all and 5=Very much.
  Higher score indicates more satisfaction. Positive change in score indicates improvement.
General Academic Self-Efficacy scale (GASE) | Baseline, Day 42, Day 84
  The GASE is a short and concise five-item measure of the longer form Academic self-efficacy (ASE) scale. The scale assesses a student's global belief in his or her ability to master the various academic challenges in an academic setting and is considered an essential antecedent of wellbeing and performance.
  Higher score indicates more self-efficacy. Positive change in score indicates improvement.
Mental Health Quality of Life Scale (MHQoL) | Baseline, Day 42, Day 84
  The MHQoL is a standardized, validated self-report measure of quality of life that has been developed for use in people with mental health problems.18 It consists of 7-items covering self-image, independence, mood, relationships, daily activities, physical health, and future measured on a 4-point Likert scale ranging from "Very satisfied" to "Very dissatisfied," and an analogue scale from regarding psychological well-being where 0 = "worst imaginable psychological well-being" and 10 = "best imaginable psychological well-being."
  Higher score indicates a better quality of life. Positive change in score indicates improvement.
Adult ADHD Self-Report Scale (ASRS) | Baseline, Day 42, Day 84
  The ASRS v1.1 is an 18-item self-report validated questionnaire designed to assess ADHD symptoms in adults. No total score or diagnostic likelihood is utilized for the twelve questions. Frequency scores are used to determine if the patient has symptoms highly consistent with ADHD in adults. The frequency-based response is more sensitive with certain questions.
  Greater frequency indicates higher symptom consistency with ADHD in adults. Negative change indicates improvement.
Patient Health Questionnaire-4 (PHQ-4) | Baseline, Day 42, Day 84
  PHQ-4 is an ultra-brief, validated screening assessment for anxiety and depression, consisting of four-items that are scored on a Likert scale of 0 (not at all), 1 (several days), 2 (more than half the days), and 3 (nearly every day).
  A higher score indicates greater levels of depression and anxiety. Negative change indicates improvement.

OTHER OUTCOMES:
System Usability Scale (SUS) | Day 84
  The SUS is a brief, validated 10-item questionnaire that is designed to evaluate a wide variety of products and services, including hardware, software, mobile devices, websites and applications.22 The SUS consists of 10 items rated on a 5-point Likert scale that range from "strongly agree" to "strongly disagree." Results interpretation typically requires normalizing the scores to produce a percentile ranking; however, a SUS score above 68 can generally be considered above average, and a score below 68, generally considered below average.

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Stamatis, PhD, Principal Investigator — Akili Interactive Labs, Inc.
Locations (2):
- United States (2):
  - Villa Maria College, Cheektowaga, New York
  - Landmark College, Putney, Vermont

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.